CLINICAL TRIAL: NCT06629441
Title: Effectiveness and Safety of Probiotics, BC99 in Relieving Anxiety and Depression in Adults
Brief Title: Effectiveness and Safety of Probiotics in Relieving Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024013
Record Dates: First submitted 2024-09-18; First posted 2024-10-08 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): 10B CFU/Sachet/Day BC99, before meals, Storage: Store in cool and dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic group
- Placebo (Placebo Comparator): Maltodextrin Sachet/Day, before meals, Storage: Store in cool and dry place without sun exposure.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Probiotic group — taking 10 billion CFU probiotic one sachet one time, lasting 56 days.
  Arms: Probiotic group
Dietary Supplement: Placebo group — taking maltodaxtrin one sachet one time, lasting 56 days.
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness and safety of probiotics in relieving anxiety and depression in adults, in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, Written, and Signed Informed Consent: Agreeing to participate in the study.
2. Ability to Complete the Study According to Protocol: Able to meet the requirements of the study protocol.
3. Age: 18-65 years old.
4. Depression and Anxiety Scores:

   * Hamilton Depression Rating Scale (HAMD-17) score of 20 or higher, or
   * Hamilton Anxiety Rating Scale (HAMA) score of 14 or higher.
5. No History of Certain Conditions: No history of heart, liver, kidney, nervous system, psychiatric disorders, or metabolic abnormalities.

Exclusion Criteria:

1. Past Diagnosis of Certain Conditions: Individuals with a history of other clearly diagnosed psychiatric disorders, intellectual disabilities, consciousness disorders, complete aphasia, bipolar disorder, treatment-resistant depression, or suicidal thoughts.
2. Pregnant or Breastfeeding Women: Individuals who are pregnant or breastfeeding.
3. Use of Certain Medications: Individuals who have used anti-anxiety, anti-depressant medications, or mood stabilizers within the past month.
4. Allergy History: Individuals with allergic constitutions or a history of drug allergies, or those with severe systemic diseases.
5. Substance Abuse History: Individuals with a history of alcohol or psychoactive substance abuse within the past 3 months.
6. Impact of Medications on Gut Microbiota: Individuals who have used medications affecting gut microbiota (including antibiotics, probiotics, mucosal protectors, traditional Chinese medicine, etc.) continuously for more than 1 week in the month prior to screening.
7. Discontinuation or Addition of Medications: Individuals who have stopped taking the study medication or started taking other medications, making it difficult to assess efficacy or with incomplete data.
8. Use of Similar Products: Individuals who have taken items similar to the study product in the short term, affecting the evaluation of results.
9. Inability to Participate: Research participants who cannot participate in the study due to personal reasons.
10. Other Exclusions: Participants deemed unsuitable for the study by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale (HAMD-17) total score from baseline to Week 8 | Baseline and Week 8
  Clinician-rated HAMD-17; higher scores indicate more severe depressive symptoms. Negative change denotes improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- The 1st Affiliated Hospital of He'nan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No